CLINICAL TRIAL: NCT03459950
Title: China Academy of Chinese Medical Sciences
Brief Title: Experimental Research Center of China Academy of Chinese Medical Sciences
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jun Song (Other)
Responsible Party: Sponsor-Investigator, Jun Song, Researcher, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: Jun Song
Record Dates: First submitted 2018-03-02; First posted 2018-03-09 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Insomnia group: 60 patients with chronic insomnia are included in the Chronic Insomnia group. Men and women half, the age of 18-60 years old, signature to the Information for Patient.
- Normal control group: 60 normal people are included in the normal control group. Men and women half, the age of 18-60 years old, signature to the Information for Patient.

SUMMARY:
Insomnia belongs to the category of"sleepless"in Chinese medicine. Sleepless is defined as a persistent sleep disorder, results in some form of daytime impairment.

Traditional Chinese medicine(TCM) has obvious advantages in the treatment of chronic insomnia, but there have some subjective and objective obstacles in the advantages of TCM treatment of replication, promotion, and popularization. Therefore, it is necessary to carry out the research from a multi-angle, and further summarize the ideas and methods from the perspective of TCM, to make it more objective, visual and standardized.

Insomnia is a clinical manifestation of the disorders of the Zang and Fu, and it can further aggravate the dysfunction of the Zang and Fu. The Traditional Chinese medicine believes that, outward is the internal manifestation. Infrared image can reflect the state of cold and heat, yin and yang in all parts of human body. So it is called the CT of TCM. Pre-study found that patients with sleep disorders have different infrared image than normal changes. Polysomnography is currently recognized as the golden indicator of sleep research. Polysomnography can monitor the whole sleep process, and study the sleep structure by the related indexes, which is a basic technique for Sleep medical research and diagnosis of sleep disorders, and a standard method of evaluating sleep-related pathophysiology and sleep architecture. We will study the relationship between sleep structure of the PSG, the characteristics of infrared image, the four diagnostic information of TCM, and the self-rating scales of sleep and psychology in patients with chronic insomnia.

DETAILED DESCRIPTION:
Insomnia is a clinical manifestation of the disorders of the Zang and Fu, and it can further aggravate the dysfunction of the Zang and Fu. The Traditional Chinese medicine believes that, outward is the internal manifestation. Infrared image can reflect the state of cold and heat, yin and yang in all parts of human body. So it is called the CT of TCM. Pre-study found that patients with sleep disorders have different infrared image than normal changes. Polysomnography is currently recognized as the golden indicator of sleep research. Polysomnography can monitor the whole sleep process, and study the sleep structure by the related indexes, which is a basic technique for Sleep medical research and diagnosis of sleep disorders, and a standard method of evaluating sleep-related pathophysiology and sleep architecture.

In order to further understand sleep disorders and improve the efficiency of Chinese medicinein treating sleep disorders. We will study the relationship between sleep structure of the PSG, the characteristics of infrared image, the four diagnostic information of TCM, and the self-rating scales of sleep and psychology in patients with chronic insomnia

ELIGIBILITY:
Chronic Insomnia group Inclusion criteria Chronic insomnia diagnosis consistent with the criteria of International Classification of Sleep Disorder, third version (ICSD-3), PSQI score is greater than 16, 18 to 60 years of age, written informed consent.

Exclusion criteria Sedative-hypnotic, antidepressant with sedative effect, atypical antipsychotic drugs that have been used in 7 days, patients with severe neurological and psychiatric disorders, with systemic immune diseases and significant skin diseases, and who is unable to test for various reasons.

Normal control group Inclusion criteria Subjects do not have chronic insomnia or insufficient of sleep near a month, normal level of blood pressure, blood sugar, and blood lipid, 18 to 60 years of age, written informed consent.

Exclusion criteria PSQI score is greater than 7, people who have been taken drugs that affect sleep in the past week, have obvious clinical symptoms of coronary heart disease and cerebrovascular disease, and have severe neurological and psychiatric disorders, systemic immune diseases, and who is unable to test for various reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 patients with sleep disorder are included in the sleep disorder group and 60 in the normal control group, men and women half, the age of 18-60 years old, signature to the Information for Patient.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Infrared image | 2019.9
  Observed subjects in various regions or regions hot △T, which is the average temperature difference between body and body surface

CONTACTS AND LOCATIONS:
Locations (1):
- Experimental Research Center of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No